CLINICAL TRIAL: NCT05009563
Title: Evaluation of COVID-19 by Whole-body FDG-PET/CT
Brief Title: COvid iMaging With POSitron Emission Tomography
Acronym: COMPOSIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Semmelweis University Department of Pulmonology (Unknown); Semmelweis University Medical Imaging Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPOSIT Study
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus Infection
Keywords: COVID19; PET-CT; brain; lung
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatients with RT-PCR proven SARS-CoV-2 infection (Experimental): Inpatients with real-time reverse-transcriptase polymerase chain reaction (RT-PCR) proven SARS-CoV-2 infection of the Department of Pulmonology of Semmelweis University who will undergo whole-body FDG-PET/CT
  Interventions: Radiation: FDG-PET/CT
- patients undergoing FDG-PET/CT for oncological indication (Active Comparator): Age- and gender-matched group of patients undergoing FDG-PET/CT for oncological indication in the same time period
  Interventions: Radiation: FDG-PET/CT

INTERVENTIONS:
Radiation: FDG-PET/CT — whole-body F-18-fluoro-deoxy-glucose positron emission tomography/computed tomography

SUMMARY:
We aim to study if metabolic intensity and extent according to pathologic pulmonary 18F-2-fluoro-2-deoxy-D-glucose (FDG)-uptake may correlate with the course of COVID-19 pneumonia and potentially yield prognostic value. Moreover, we aim to assess permanent changes after Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, such as pulmonary fibrosis and neuropsychiatric symptoms (anosmia, depression, fatigue) where evaluation with FDG-positron emission tomography (PET/CT) might have an impact on further patient care.

DETAILED DESCRIPTION:
Several case studies confirmed increased FDG-uptake on PET scans corresponding to typical pulmonary lesions on chest CT scans in patients with COVID-19 pneumonia. Furthermore, increased FDG-uptake most likely caused by inflammatory changes in SARS-CoV-2 infection were described in other organs, such as mediastinal lymph nodes, bone marrow, and the spleen. As COVID-19 frequently presents with anosmia and on rare occasions, symptoms of encephalitis, metabolic changes in the central nervous system (CNS) were also investigated by FDG-PET/CT, showing hypometabolism in the olfactory gyrus and the limbic system, while hypermetabolism was observed in the basal ganglia and the cerebellar vermis. Late changes in pulmonary CT-morphology, most commonly interstitial thickening and crazy paving are observed, suggesting permanent lung damage after SARS-CoV-2 infection in certain cases. Evaluation of metabolic activity of acute and late inflammatory changes could potentially provide clinical benefit as dedicated medication could be started to prevent further organ damage due to prolonged inflammation.

We aim to evaluate metabolic alterations in the lung parenchyma and potential extrapulmonary locations related to to COVID-19 with FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with RT-PCR proven SARS-CoV-2 infection of the Department of Pulmonology of Semmelweis University

Exclusion Criteria:

* Age<40 years for men and <45 years for women
* Pregnancy
* Clinically unstable patients
* Patients in need of mechanical ventilation support
* Patients with known malignant disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-01-04 (Estimated); Study Completion 2022-01-04 (Estimated)

PRIMARY OUTCOMES:
extrapulmonary increased FDG-uptake | 3 months
  observation of sites with extrapulmonary hypermetabolic foci in possible conjunction with COVID-19 and brain metabolic changes, with follow-up scan

SECONDARY OUTCOMES:
total pulmonary metabolic inflammatory volume | 3 months
  measurement of metabolic activity of COVID-19 pneumonia and changes on follow-up scan

OTHER OUTCOMES:
cognitive status and quality of life | 3 months
  investigation of possible COVID-19-related cognitive changes and impact on quality of life, with follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pál Maurovich Horvat, MD PhD MPH, Principal Investigator — Semmelweis University Medical Imaging Centre
Locations (1):
- Semmelweis University Medical Imaging Centre, Budapest, Pest County, Hungary

REFERENCES:
- [Background] Qin C, Liu F, Yen TC, Lan X. 18F-FDG PET/CT findings of COVID-19: a series of four highly suspected cases. Eur J Nucl Med Mol Imaging. 2020 May;47(5):1281-1286. doi: 10.1007/s00259-020-04734-w. Epub 2020 Feb 22. PMID 32088847
- [Background] Zou S, Zhu X. FDG PET/CT of COVID-19. Radiology. 2020 Aug;296(2):E118. doi: 10.1148/radiol.2020200770. Epub 2020 Mar 6. No abstract available. PMID 32142399
- [Background] Liu C, Zhou J, Xia L, Cheng X, Lu D. 18F-FDG PET/CT and Serial Chest CT Findings in a COVID-19 Patient With Dynamic Clinical Characteristics in Different Period. Clin Nucl Med. 2020 Jun;45(6):495-496. doi: 10.1097/RLU.0000000000003068. PMID 32332319
- [Background] Cabrera Villegas A, Romero Robles LG, Boulvard Chollet XLE, Albornoz Almada MC, Mangas Losada M, Garrastachu P, Canete Sanchez FM, Ramirez Lasanta R, Delgado Bolton RC. [18F]-FDG PET/CT in oncologic patients with unsuspected asymptomatic infection with SARS-CoV-2. Eur J Nucl Med Mol Imaging. 2021 Mar;48(3):786-793. doi: 10.1007/s00259-020-04979-5. Epub 2020 Sep 16. PMID 32936372
- [Background] Dietz M, Chironi G, Claessens YE, Farhad RL, Rouquette I, Serrano B, Nataf V, Hugonnet F, Paulmier B, Berthier F, Keita-Perse O, Giammarile F, Perrin C, Faraggi M; MONACOVID Group. COVID-19 pneumonia: relationship between inflammation assessed by whole-body FDG PET/CT and short-term clinical outcome. Eur J Nucl Med Mol Imaging. 2021 Jan;48(1):260-268. doi: 10.1007/s00259-020-04968-8. Epub 2020 Jul 25. PMID 32712702
- [Background] Guedj E, Million M, Dudouet P, Tissot-Dupont H, Bregeon F, Cammilleri S, Raoult D. 18F-FDG brain PET hypometabolism in post-SARS-CoV-2 infection: substrate for persistent/delayed disorders? Eur J Nucl Med Mol Imaging. 2021 Feb;48(2):592-595. doi: 10.1007/s00259-020-04973-x. Epub 2020 Jul 30. PMID 32728799
- [Background] Grimaldi S, Lagarde S, Harle JR, Boucraut J, Guedj E. Autoimmune Encephalitis Concomitant with SARS-CoV-2 Infection: Insight from 18F-FDG PET Imaging and Neuronal Autoantibodies. J Nucl Med. 2020 Dec;61(12):1726-1729. doi: 10.2967/jnumed.120.249292. Epub 2020 Jul 24. PMID 32709734
- [Background] Yu M, Liu Y, Xu D, Zhang R, Lan L, Xu H. Prediction of the Development of Pulmonary Fibrosis Using Serial Thin-Section CT and Clinical Features in Patients Discharged after Treatment for COVID-19 Pneumonia. Korean J Radiol. 2020 Jun;21(6):746-755. doi: 10.3348/kjr.2020.0215. PMID 32410413
- [Background] Wang Y, Dong C, Hu Y, Li C, Ren Q, Zhang X, Shi H, Zhou M. Temporal Changes of CT Findings in 90 Patients with COVID-19 Pneumonia: A Longitudinal Study. Radiology. 2020 Aug;296(2):E55-E64. doi: 10.1148/radiol.2020200843. Epub 2020 Mar 19. PMID 32191587